CLINICAL TRIAL: NCT04470700
Title: Predictors of Delay in Treatment of Urinary Incontinence Among Pakistani Women - a Cross-sectional Study
Brief Title: Predictors of Delay in Treatment of Urinary Incontinence
Acronym: Predictors
Status: Completed | Type: Observational
Sponsor: Shazia Saaqib (Other)
Responsible Party: Sponsor-Investigator, Shazia Saaqib, Assistant Professor Obstetrics and Gynecology, King Edward Medical University
Organization: King Edward Medical University (Other)
Other Study IDs: 711/RC/KEMU
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- subjects with greater than 3years delay: Subjects with delay in treatment of Urinary incontinence greater than three years
- subjects with less than three years delay: Subjects with delay in treatment of Urinary incontinence lesser than three years

SUMMARY:
246 women were selected as participants to fill and submit the Study Proforma among 264 incontinent women. The Performa included demographic features of the subjects, their chronic ailments, psychosocial effects, reasons for the delay, and Incontinence Questionnaire UI-short form of incontinence characteristics. We selected a sample of 198 completed questionnaires to be included in the study. IBM spss statistics 20(SPSS Inc, Chicago, IL, USA) were used to find predictors of delay in treating urinary incontinence.

DETAILED DESCRIPTION:
Study design and participants:

A cross-sectional survey of 198 women with incontinence was conducted at lady Willingdon hospital from June 1, 2019, to November 30, 2020. The medical officers of gynecology outdoor scrutinized all the women who had complained of urinary incontinence for at least one year and did not previously pursue any treatment for this problem.

246 participants who fulfilled the study criteria signed written informed consent and got their Proforma filled either by themselves or by assisting the medical officer.

In previous studies, delay to the treatment of >3 years was considered significant; thus, all eligible women were divided into two groups based on the delay of up to three years and more than 3 years according to the duration of incontinence as stated by the subject and studied for predictors of incontinence.

Ethical approval This study had ethical approval from King Edward Medical University, Pakistan. the study was conducted according to the Declaration of the Helsinki and obtained informed consent from participants before the study commenced. All information collected from the participants was kept confidential, and Proformas were kept in a file in the custody of the main investigator after entering data in the spss datasheet.

Statistical analysis. The study results were calculated with SPSS version 20 (SPSS Inc., Chicago, IL, USA). The means and standard deviation were used to calculate the age of subjects and the duration of delay in seeking treatment. The subjects with potential risk factors were represented as numbers and percentages. The subjects with a short delay(less than or equal to three years) and a long delay (greater than three years) were presented as numbers and percentages for reporting their incontinence. Univariate analysis was performed on all risk factors of delay and then multivariate analysis on significant risk factors to determine the most commonly shared factors for delay in seeking treatment. P-value ≤ 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* The women who had the complaint of urinary incontinence for at least one year and did not pursue any treatment for this problem previously.
* age greater than 18 years
* urinary leakage for once a week during the previous three months.
* Incontinent women with or without chronic medical problems

Exclusion Criteria:

* urinary tract infection
* patients with pregnancy or within three months postpartum
* severe mental illness (unable to answer the questionnaire correctly)
* terminal stage illness (liver disease, kidney disease, or malignancy)

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female subjects above18 years of age
Study Population: The women who had complained of urinary incontinence for at least one year and did not pursue any treatment for this problem previously.
Sampling Method: Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Predictors of delay in treatment of urinary incontinence | 6months from1st june2019 to 30 november 2019
  the risk factors of incontinence treatment delay wich are shared by the women with delayed help seeking behaviour

CONTACTS AND LOCATIONS:
Overall Officials: Shazia Saaqib, FCPS,MCPS, Study Chair — King Edward Medical University,Lahore, Pakistan
Locations (1):
- Lady Willingdon Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
The data will be shared after publication on a reasonable request.

REFERENCES:
- [Result] Sensoy N, Dogan N, Ozek B, Karaaslan L. Urinary incontinence in women: prevalence rates, risk factors and impact on quality of life. Pak J Med Sci. 2013 May;29(3):818-22. doi: 10.12669/pjms.293.3404. PMID 24353635
- [Result] Norton PA, MacDonald LD, Sedgwick PM, Stanton SL. Distress and delay associated with urinary incontinence, frequency, and urgency in women. BMJ. 1988 Nov 5;297(6657):1187-9. doi: 10.1136/bmj.297.6657.1187. No abstract available. PMID 3144344
- [Result] Corcos J, Gajewski J, Heritz D, Patrick A, Reid I, Schick E, Stothers L; Canadian Urological Association. Canadian Urological Association guidelines on urinary incontinence. Can J Urol. 2006 Jun;13(3):3127-38. PMID 16813704
- [Result] Lasserre A, Pelat C, Gueroult V, Hanslik T, Chartier-Kastler E, Blanchon T, Ciofu C, Montefiore ED, Alvarez FP, Bloch J. Urinary incontinence in French women: prevalence, risk factors, and impact on quality of life. Eur Urol. 2009 Jul;56(1):177-83. doi: 10.1016/j.eururo.2009.04.006. Epub 2009 Apr 10. PMID 19376639
- See also: The Prevalence and Determinants of Health Care-Seeking Behavior for Urinary Incontinence in United Arab Emirates Women — https://doi.org/10.1007/s001920050038
- See also: The Relationship Between Urinary Incontinence, Mobility Limitations, and Disability in Older Women — https://doi.org/10.1007/s13670-017-0202-4